CLINICAL TRIAL: NCT00401102
Title: An Open-clinical Trial of Interpersonal Psychotherapy for Depressed Adolescents (IPT-A) for Depressed Adolescents Engaged in Non-suicidal Self-injury
Brief Title: Interpersonal Psychotherapy for Depressed Adolescents Engaging in Non-suicidal Self-injury
Acronym: IPT-ASI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: MINT: Mental Health Initiative (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5332
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2012-12

CONDITIONS: Depression; Self-injurious Behavior
Keywords: self-injurious behavior; depression; adolescents; psychotherapy
MeSH Terms: conditions — Depression; Self-Injurious Behavior | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interpersonal psychotherapy (Other): All participants received interpersonal psychotherapy adapted for self-injury
  Interventions: Behavioral: Interpersonal Psychotherapy for Depressed Adolescents

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Depressed Adolescents — Open clinical trial of IPT-ASI for depressed and self-injuring adolescents, 12-18 years. Goal is to assess feasibility of using IPT-A protocol for teens with co-morbid depression and self-injury. All eligible participants receive 12 weeks of individual IPT-ASI with optional monthly booster sessions. IPT-ASI is a psychosocial intervention that focuses on the importance of interpersonal relationships in relation to psychological functioning. The first phase (4 weeks) includes a review of depression and self-injury symptoms, psycho-education about depression and self-injury, and a detailed assessment of the patient's important interpersonal relationships. The middle phase (weeks 5-9) involves interpersonal skill building, including communication skills, affect identification and expression, problem solving. The final phase ( weeks 10-12) involves review of skills, generalization of skills to other relationships, termination.

SUMMARY:
The purpose of this study is to examine the feasibility of using Interpersonal Psychotherapy for Depressed Adolescents (IPT-A) to treat adolescents who are experiencing symptoms of depression and are engaging in non-suicidal self-injurious behaviors. The trial will include recruiting 10 particpants, administering 12-sessions of individual IPT-A, and determining how the IPT-A protocol needs to be amended to adequately address the self-injury in addition to depression.

DETAILED DESCRIPTION:
Engagement in non-suicidal self-injury (NSSI), purposefully harming oneself without the conscious intent to die such as cutting or burning, is pervasive among adolescents. Lifetime prevalence estimates among community samples of high school students range from 13.0% to 23.2%. Despite the significance of this public health problem, there are no known interventions that successfully reduce the frequency of NSSI or prevent NSSI in adolescents. The goal of the current study is to develop an effective psychosocial intervention for NSSI among adolescents who are engaging in self-injury and have a depressive disorder. Specifically, we will amend Interpersonal Psychotherapy for Depressed Adolescents (IPT-A), a psychotherapy that has demonstrated efficacy in treating depressed adolescents (Mufson et al., 1994, 1999, 2004), for use with adolescents with depression who are engaging in NSSI, with the ultimate goal of curing the depression and NSSI. Ten participants will be administered IPT-A and assessed several times throughout the course of the trial. It is expected that IPT-A will be a useful treatment for co-morbid depression and self-injury, although adaptations to the protocol will likely be needed to address the behavioral aspect of the self-injury. Data analyses will be descriptive in nature and involve examining the individual trajectories of depression and NSSI over time. The data obtained from the current study will lay the groundwork for an ultimate randomized controlled trial in which we plan to compare IPT-A versus nondirective supportive therapy in the treatment of co-morbid depression and NSSI.

ELIGIBILITY:
Inclusion Criteria:

1. 12 to 18 years of age
2. Diagnosis of MDD, Dysthymic Disorder, Depressive Disorder NOS, Adjustment Disorder with depressed Mood
3. Non-suicidal self-injurious behavior
4. CDRS >= 36
5. C-GAS <= 65
6. English speaking patient
7. One English speaking caregiver -

Exclusion Criteria:

1. Suicide attempt within past 6 months or actively suicidal
2. Severe incident of non-suicidal self-injury in past 3 months
3. Severe episode of MDD
4. Treatment resistant non-suicidal self-injury
5. Frequent non-suicidal self-injury
6. Mentally retarded
7. Current diagnosis of: PTSD, OCD, Schizophrenia, Bipolar Disorder, Psychosis, Substance Dependence, ADHD
8. Current substance use
9. Currently in active treatment for same condition
10. Currently taking antidepressant medication
11. Medical illness likely to interfere with treatment -

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2006-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Jacobson, PhD, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: All participants recieved Interpersonal psychotherapy
Period: Overall Study
Arm/Group | Group 1
Started | 12
Completed | 5
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: CGI
Time Frame: 1 week
Reporting Status: Not Posted

2. Primary Outcome: C-GAS
Time Frame: 1 month
Reporting Status: Not Posted

3. Primary Outcome: CDRS
Time Frame: 1 week
Reporting Status: Not Posted

4. Primary Outcome: Self-Injurious Thoughts and Behaviors Interview
Time Frame: 8 weeks
Population: Data for all subjects who completed the study was examined - however because this was a small pilot study and only 5 subjects completed treatment, no statistical tests were completed.
Measure: Mean (Standard Deviation); unit: episodes of self-injury past month
Arm/Group | Group 1
Number analyzed (Participants) | 5
episodes of self-injury past month | 0.4 (0.9)

5. Primary Outcome: Self-injury Monitoring Card
Time Frame: 1 month
Reporting Status: Not Posted

6. Secondary Outcome: Beck Depression Inventory
Time Frame: 2 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Multidimensional Anxiety Scale for Children
Time Frame: recently
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No